CLINICAL TRIAL: NCT05757674
Title: Analysis of the Intestinal Microbiome in Patients With Wet Age-related Macular Degeneration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Andreas Katsanos, Associate Professor of Ophthalmology, University of Ioannina
Other Study IDs: 20(7)-15/4/2020.
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients
  Interventions: Other: Sample examination
- Control: Control
  Interventions: Other: Sample examination

INTERVENTIONS:
Other: Sample examination — No intervention will be performed

SUMMARY:
Analysis of the Intestinal Microbiome in Patients With Wet Age-related Macular Degeneration

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed neovascular age-related macular degeneration.

Exclusion Criteria:

* Chronic gastrointestinal disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed patients with neovascular age-related macular degeneration from the area of North-West Greece
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Intestinal microbiome profile | 2022-2023
  Intestinal microbiome profile

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: Undecided